CLINICAL TRIAL: NCT04405726
Title: Study of Clinical, Biological and Genetic Prognostic Factors of SARS-CoV-2 Infection in Patients Admitted in the Strasbourg University Hospitals
Brief Title: Prognostic Factors of COVID19
Acronym: Covid-HUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7760
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-05

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; Covid-19; Prognostic factors; Genetic factors; T and B cell immune response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is an emerging disease, for which no specific treatment options are currently available. Since the end of February 2020, and due to a SARS-CoV-2 superspreading event (religious meeting), the Strasbourg University Hospital (HUS) had faced a sudden increase of the number of COVID-19-positive patients in serious condition requiring hospitalization. At the same time, many people develop only mild or moderate symptoms. To date, the prognostic factors for the course of SARS-CoV-2 infection are unknown. The primary purpose of the "COVID-HUS" protocol is to investigate viral and host-related factors to understand the pathophysiology of COVID infection and to open the way for new diagnostic, prognostic and therapeutic strategies against SARS CoV-2 .

The secondary objectives are

* Monitoring of viral replication of SARS-CoV-2 in the blood and respiratory tract in infected patients
* Monitoring of the humoral and cellular response directed against SARS-CoV-2
* Identification of factors leading to significant and / or prolonged viral replication of SARS-CoV-2 in the blood or respiratory samples
* Evaluation of the benefit of possible treatments implemented following the diagnosis of SARS-CoV-2 infection
* Exploration of the B and T immune repertoire sequences targeting SARS-CoV-2 in infected patients
* Typing of the HLA system in infected patients

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric with suspicion or a confirmed SARS-CoV-2 infection
* Patient who has signed a non-opposition form (or a form signed by a family member or a support person if the seriousness of the patient's condition and the emergency situation do not allow it) or who has given his oral agreement to the doctor

Exclusion Criteria:

* Patient's explicit refusal to participate
* Subject deprived of liberty or subject to the protection of justice
* Subject under guardianship or trusteeship

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric with suspicion or a confirmed SARS-CoV-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-27 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Clinical Presentation and Incidence of Covid-19 Infection in patients hospitalised in Strasbourg Hospital | From 1st March 2020 to 1st March 2021

CONTACTS AND LOCATIONS:
Overall Officials: Samira FAFI-KREMER, PharmD, PhD, Study Director — Laboratoire de Virologie Plateau Technique de Microbiologie
Locations (1):
- Service de Virologie - Hôpital Civil, Strasbourg, France

REFERENCES:
- [Derived] Partouche N, Maumy M, Chamaraux-Tran TN, Bertrand F, Schneider F, Meyer N, Solis M, Fafi-Kremer S, Noll E, Pottecher J. Does the IL-6/KL-6 ratio distinguish different phenotypes in COVID-19 Acute Respiratory Distress Syndrome? An observational study stemmed from prospectively derived clinical, biological, and computed tomographic data. PLoS One. 2025 May 21;20(5):e0321533. doi: 10.1371/journal.pone.0321533. eCollection 2025. PMID 40397955
- [Derived] Gallais F, Velay A, Nazon C, Wendling MJ, Partisani M, Sibilia J, Candon S, Fafi-Kremer S. Intrafamilial Exposure to SARS-CoV-2 Associated with Cellular Immune Response without Seroconversion, France. Emerg Infect Dis. 2021 Jan;27(1):113-21. doi: 10.3201/eid2701.203611. Epub 2020 Dec 1. PMID 33261718